CLINICAL TRIAL: NCT01963572
Title: A Continuing Cancer Service Model Emphasizing on Functional Restoration: Model for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201212092RINC; NSC 102-2314-B-002-030-MY3
Record Dates: First submitted 2013-10-06; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Quality of Life
Keywords: Breast cancer; Care model; Physical Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- surveillance group (SG) (Experimental): SG will have health education brochure and free class from the first visit post-operatively but CG will only have the brochure. Moreover, SG will be screened every time when they visit the clinics. If there is any early sign of impairment, professional advice and counseling will be given additionally.
  Interventions: Other: SG will be screened every time when they visit the clinics.
- general care group (CG) (No Intervention): CG raises any health-related question, they can be answered.

INTERVENTIONS:
Other: SG will be screened every time when they visit the clinics.
  Arms: surveillance group (SG)

SUMMARY:
Background and Purposes: Cancer is the leading cause of our mortality. It threatens people's life and quality of life (QOL). Although the incidence of cancer is still rising, with the promotion of cancer screening and progression of medical technology, its survival rate is improving. However, the sequels from cancer or its treatment and the side effects impact the patients along with their lives. Breast cancer is the most incident cancer in women with high survival rate, continuing care after the diagnosis and treatment is much more needed. This study is using breast cancer as an example to establish a continuing service model. This study aims (1) to establish a tailored, continuing care model which emphasizes on breast cancer patients' function. (2) To investigate the effectiveness of the new care model comparing with the control. (3) To find a cutting point of bioelectrical impedance to identify late development of lymphedema.

Methods: This is a randomized-controlled trial expanding for 3 years. Women being newly diagnosed with breast cancer and first OPD visit after operation at National Taiwan University Hospital will be invited to join the surveillance and care system. Exclusion criteria are: younger than 20 years old, stage IV, recurrent or both sides involved, with other cancer diagnosis, functional impairments from previous injury or operation on the affected upper extremity and other physical or mental problem to influence the test or filling the questionnaire. It is estimated there will be 100 subjects participate this study every year. After the initial evaluation, they will be randomly allocated to surveillance group (SG) or general care group (CG). Totally, in this three-year study, there will be 200 subjects (100/group), follow-up for 0.5 to 2 years. SG will have health education brochure and free class from the first visit post-operatively but CG will only have the brochure. Moreover, SG will be screened every time when they visit the clinics. If there is any early sign of impairment, professional advice and counseling will be given additionally. In these visits, if CG raises any health-related question, they can be answered. Detailed physical examination to identify their impairments and QOL are at 3, 6, 12, 18, 24 months after operation for both groups. Patients' characteristics, functional status, QOL will be presented by descriptive statistics. T-test/Mann-Whitney U test will be used to compare the differences between patients in two groups. Survival analysis and log-rank test will be used to show the prevalence of various functional impairments and test their difference. ROC curve will be used to find the cutting point for prediction of lymphedema.

Expected Results: It is expected (1) to set up the education program and brochure for breast cancer patients. (2) to establish a continuing surveillance and care model for breast cancer patients and extending to all cancers. (3) Women in the new care model will have less impairment and higher QOL comparing with women at the same post-operative stage. (4) To find out the prevalence of functional impairments from the data of control group. (5) A cutting point of bioelectrical impedance to identify late development of lymphedema will be found. (6) To train the team members of cancer care and research.

ELIGIBILITY:
Inclusion Criteria:

* Women being newly diagnosed with breast cancer and first OPD visit after operation at National Taiwan University Hospital will be invited to join the surveillance and care system

Exclusion Criteria:

* Younger than 20 years old, stage IV, recurrent or both sides involved, with other cancer diagnosis, functional impairments from previous injury or operation on the affected upper extremity and other physical or mental problem to influence the test or filling the questionnaire.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
prevalence of body impairments | 2 years
  Standard physical examination including body composition, arm circumferences, shoulder range of motion and strength, grip strength, muscle length, posture, pain assessment will be performed at baseline and 5 time points of follow-up for both groups for detecting any kind of body impairment.
changes of functional status | baseline, 3,6,12,18 and 24 months
  several self-administrated questionnaires including ECOG, DASH, EORTC QLQ-C30, CFS, HADS will be used for assessing changes of functional status from baseline and 5 time points of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Principal Investigator — Gratuate School of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan
Locations (1):
- Graduate Scahool of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan